CLINICAL TRIAL: NCT02376855
Title: A Study of the Implementation of an Electronic Consultation ("eConsult") Platform to Increase Specialist Access for Patients in Underserved Populations: Impact on Provider Experience, Wait Times and Cost
Brief Title: A Study of the Implementation of an Electronic Consultation ("eConsult") Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Health Center, Inc. (Industry)
Collaborators: Connecticut Health Foundation (Other); University of Connecticut (Other); UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1023
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Diseases
Keywords: Health Services Accessibility
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Providers in the Control group followed standard care protocols. If they deemed a patient was in need of cardiology consultation, a referral was created using the standard process. The referral was processed by a referral coordinator and transmitted to an appropriate cardiologist. An appointment was then scheduled for the patient to have an in-person consultation with a cardiologist.
- eConsult (Experimental): The intervention consisted of an eConsult pathway and standardized protocol for PCPs to obtain cardiology consults using a secure messaging "peer to peer" (P2P) module embedded within the EHR. Intervention providers were asked to send all cardiology referrals for their adult patients through the eConsult system. Providers could bypass the eConsult pathway for patients with established relationships with a cardiologist or for whom providers felt a consult was urgent (required a face-to-face visit within a week or less). eConsults contain reason for consult, relevant test results, records or reports but are sent electronically to a Cardiology Consultant for review. eConsults were responded to within two business days. Responses were case-specific and generally contained recommendations for management, additional testing, or a face-to-face cardiology visit. The PCP was responsible for considering/acting upon recommendations and determining when an eConsult was complete.
  Interventions: Other: eConsult

INTERVENTIONS:
Other: eConsult — An electronic consultation or "eConsult" is a secure message consult that allows specialists to provide advice on cases without seeing a patient face to face. They contain a reason for consult, any relevant tests, procedures or reports. The responsibility lies with the primary care provider to act, or not act on the advice as they deem fit.
  Arms: eConsult

SUMMARY:
The purpose of this study is to evaluate the implementation of an electronic consultation model for specialty services (eConsults) to improve quality of care and reduce health system costs. An eConsult is a non-face-to-face consultation between a primary care provider and a specialist that takes place via secure messaging.

DETAILED DESCRIPTION:
The study is a randomized, controlled trial where the intervention is the evidence-based eConsult model in which consults are submitted by electronic, secure messaging to a specialist for review and "virtual" consultation. Primary Care Providers will be randomized to the control or intervention group. In the intervention group, ALL new, non urgent, adult cardiology referrals will be submitted to the eConsult Cardiology team for an eConsult. Consults for children (age <18) and consults for patients who already have an established relationship with another cardiologist will not be eligible for an eConsult. Urgent consults, such as those for patients with active chest pain or other acute conditions, will not be submitted for eConsult and should instead be handled by the on-site care team as per the standard protocol. For eConsults, the consult will be submitted using the eConsult pathway within the electronic health record. eConsults will be created in the same way that standard referrals are created, with attachment of a treatment summary, EKG, relevant results, and specification of the consultative question. The eConsult will be received by the intervention Cardiology team and reviewed within 2 business days. One cardiologist per day will be assigned to review and respond to eConsults.

The result will be received by the primary care provider who will be responsible for acting appropriately on the cardiologist's recommendations. Recommendations will be case specific and may include one of three broad areas of suggestion: 1) suggestions for ongoing management by the primary care provider, 2) suggestions for additional testing in advance of a cardiology face to face appointment or to better determine a next course of action, and 3) immediate cardiology referral.

For each of these options, the primary care provider will be responsible for following up and implementing the recommendations made by the Cardiologist. When referral is recommended the primary care provider will refer the patient to the cardiologist of their choice based on their location and the patient's preference. While not required, they may refer the patient to the eConsult cardiology team at University of Connecticut for face to face care if desirable, but may also refer to other Cardiologists. The intervention will last one year. Providers randomized to the control group will provide standard care which involves a traditional referral for an in-person cardiology visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care Provider at Community Health Center, Inc who work at least 30 hours per week and see adult patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time to first contact with a cardiologist | 18 months
  For eConsults, time to first contact is the time between the generation of the eConsults and when the Cardiologist replies to the eConsults. For traditional referrals, first contact is the time between the creation of the appointment and the in-person Cardiology visi.

SECONDARY OUTCOMES:
Completion of referrals | 18 months
  The percent of referrals in each group that reached completion
Adverse events | 18 months
  Adverse cardiology events, including MI, following cardiology eConsult or referral
Hospital and Emergency Department Utilization | 18 months
  Use of the hospital or Emergency Department for a cardiology complaint following an eConsult or referral
Provider Satisfaction (survey) | Baseline, 6 months, 12 months
  A survey was administered to participants to measure their satisfaction with eConsults and/or the current referral process
Number of in-person cardiology visits | 18 months
  The number of traditional, control referrals and eConsults that resulted in an in-person consultation with a cardiologist.
Total Cost Per Patient | 6 months pre and 6 months post intervention
  Clinical costs per patient in control and intervention group from claims data

CONTACTS AND LOCATIONS:
Overall Officials: J. Nwando Olayiwola, MD, MPH, Principal Investigator — Center for Excellence in Primary Care, University of California, San Francisco; Daren Anderson, MD, Principal Investigator — Weitzman Institute, Community Health Center, Inc
Locations (1):
- Community Health Center, Inc, Middletown, Connecticut, United States

REFERENCES:
- [Background] Chen AH, Yee HF Jr. Improving primary care-specialty care communication: lessons from San Francisco's safety net: comment on "Referral and consultation communication between primary care and specialist physicians". Arch Intern Med. 2011 Jan 10;171(1):65-7. doi: 10.1001/archinternmed.2010.484. No abstract available. PMID 21220663
- [Background] Yee HF Jr. The patient-centered medical home neighbor: A subspecialty physician's view. Ann Intern Med. 2011 Jan 4;154(1):63-4. doi: 10.7326/0003-4819-154-1-201101040-00011. PMID 21200042
- [Background] Chen AH, Kushel MB, Grumbach K, Yee HF Jr. Practice profile. A safety-net system gains efficiencies through 'eReferrals' to specialists. Health Aff (Millwood). 2010 May;29(5):969-71. doi: 10.1377/hlthaff.2010.0027. No abstract available. PMID 20439891
- [Background] Foy R, Hempel S, Rubenstein L, Suttorp M, Seelig M, Shanman R, Shekelle PG. Meta-analysis: effect of interactive communication between collaborating primary care physicians and specialists. Ann Intern Med. 2010 Feb 16;152(4):247-58. doi: 10.7326/0003-4819-152-4-201002160-00010. PMID 20157139
- [Background] Kim Y, Chen AH, Keith E, Yee HF Jr, Kushel MB. Not perfect, but better: primary care providers' experiences with electronic referrals in a safety net health system. J Gen Intern Med. 2009 May;24(5):614-9. doi: 10.1007/s11606-009-0955-3. Epub 2009 Mar 24. PMID 19308334
- [Background] Kim-Hwang JE, Chen AH, Bell DS, Guzman D, Yee HF Jr, Kushel MB. Evaluating electronic referrals for specialty care at a public hospital. J Gen Intern Med. 2010 Oct;25(10):1123-8. doi: 10.1007/s11606-010-1402-1. Epub 2010 May 29. PMID 20512531
- [Background] Katz MH. Golden gate to health care for all? San Francisco's new universal-access program. N Engl J Med. 2008 Jan 24;358(4):327-9. doi: 10.1056/NEJMp0706590. No abstract available. PMID 18216352
- [Background] Bindman AB, Chen A, Fraser JS, Yee HF Jr, Ofman D. Healthcare reform with a safety net: lessons from San Francisco. Am J Manag Care. 2009 Oct;15(10):747-50. PMID 19845426
- [Background] Weiner M, El Hoyek G, Wang L, Dexter PR, Zerr AD, Perkins AJ, James F, Juneja R. A web-based generalist-specialist system to improve scheduling of outpatient specialty consultations in an academic center. J Gen Intern Med. 2009 Jun;24(6):710-5. doi: 10.1007/s11606-009-0971-3. Epub 2009 Apr 15. PMID 19367375
- [Background] Fischer BS, Martinez E, Driscoll M, Conway T. Practice profile. Chicago: using evidence-based rules to make smarter referrals. Health Aff (Millwood). 2010 May;29(5):972-5. doi: 10.1377/hlthaff.2010.0068. No abstract available. PMID 20439892